CLINICAL TRIAL: NCT04628871
Title: Long-Term Follow-up of Subjects Who Were Treated With SB-318, SB-913, or SB-FIX, for Targeted Genome Editing Into the Albumin Gene in the Liver
Brief Title: Long Term Follow-up (LTFU) of Subjects Who Received SB-318, SB-913, or SB-FIX
Acronym: LTFU
Status: Active, not recruiting | Type: Observational
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-IVPRP-LT01
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia B; Mucopolysaccharidosis I; Mucopolysaccharidosis II
Keywords: Mucopolysaccharidosis I; Hurler-Scheie Syndrome; Mucopolysaccharidosis II; Hunter Syndrome; Gene Editing; Gene Therapy; Zinc Finger; SB-318; SB-913; SB-FIX; Rare; Genetic; DNA; Sangamo; ZFN; Long Term; Hemophilia B; MPS
MeSH Terms: conditions — Hemophilia B; Mucopolysaccharidosis I; Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subjects who received SB-318: Subjects who received SB-318 in clinical study SB-318-1502
  Interventions: Biological: SB-318
- Subjects who received SB-913: Subjects who received SB-913 in clinical study SB-913-1602.
  Interventions: Biological: SB-913
- Subjects who received SB-FIX: Subjects who received SB-FIX in clinical study SB-FIX
  Interventions: Biological: SB-FIX

INTERVENTIONS:
Biological: SB-318 — No study drug is administered in this study. Subject who received SB-318 in a previous trial will be evaluated in this trial for long-term safety.
  Groups: Subjects who received SB-318
Biological: SB-913 — No study drug is administered in this study. Subject who received SB-913 in a previous trial will be evaluated in this trial for long-term safety.
  Groups: Subjects who received SB-913
Biological: SB-FIX — No study drug is administered in this study. Subject who received SB-FIX in a previous trial will be evaluated in this trial for long-term safety.
  Groups: Subjects who received SB-FIX

SUMMARY:
Long-term follow-up of subjects who received SB-318, SB-913, or SB-FIX in a previous trial and completed at least 52 weeks post-infusion follow-up in their primary protocol. Enrolled subjects will be followed for a total of up to 10 years following exposure to SB-318, SB-913, or SB-FIX.

DETAILED DESCRIPTION:
Non-interventional, multi-center, long-term follow-up (LTFU) study of subjects dosed with SB-318 in the clinical study SB-318-1502, SB-913 in the clinical study SB-913-1602, and SB-FIX in clinical study SB-FIX-1501. All subjects dosed in the studies and completed at least 52 weeks post-infusion follow-up in their primary protocol will be offered to participate. Subjects who enroll will be monitored for a total of up to 10 years following exposure to the respective investigational products.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who received SB-318 under Study Protocol SB-318-1502, SB-913 under Study Protocol SB-913-1602, or SB-FIX under Study Protocol SB-FIX-1501
2. Subjects who have provided consent to participate in the LTFU study.

Exclusion Criteria:

1. Unable to comply with study visit schedule or study visit procedures.
2. Any other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have received SB-318 in Study Protocol SB-318-1502, SB-913 in Study Protocol SB-913-1602 or SB-FIX in Study Protocol SB-FIX-1501 and who have consented to participate in this Long Term Follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Long-term safety | 10 years
  Long-term safety of SB-318, SB-913, and SB-FIX by assessment of any newly-diagnosed or worsening of existing medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Sangamo Therapeutics
Locations (5):
- United States (5):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - New York University Grossman School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio